CLINICAL TRIAL: NCT02430519
Title: Effect of Autologous Platelet Rich Fibrin In Human Mandibular Molar Grade II Furcation Defects- A Clinical and Radiological Study
Brief Title: Benefits of Platelet Rich Fibrin In Mandibular Molar Furcation Defects
Acronym: PRFMMFD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr.Syed Asimuddin (Other)
Responsible Party: Sponsor-Investigator, Dr.Syed Asimuddin, Post Graduate, Panineeya Mahavidyalaya Institute of Dental Sciences & Research Centre
Organization: Panineeya Mahavidyalaya Institute of Dental Sciences & Research Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11/98/12
Record Dates: First submitted 2015-04-18; First posted 2015-04-30 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Chronic Periodontitis
Keywords: Chronic Periodontitis; Clinical Parameters; Furcation defects; Radiographic bone fill
MeSH Terms: conditions — Chronic Periodontitis; Furcation Defects | interventions — Prolactin-Releasing Hormone; Transplantation, Homologous; Guided Tissue Regeneration

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, parallel arm, interventional trial
Who Masked: Participant, Investigator
Masking Description: The eligible samples were screened and randomly assigned by lottery method by investigator KRR into PRF (Group A) and GTR + Allograft (Group B). The treatment was performed by investigator SA who was blinded to the randomization process
Oversight: Data Monitoring Committee: No

ARMS (2):
- 11 Patients with Grade II Manibular Molar Furcation (Experimental): Group A- Furcation Treatment with PRF
  Interventions: Procedure: Furcation treatment with PRF; Device: autologous platelet-rich fibrin
- 11 Patients with Grade II Mandibular Molar Furcation D (Experimental): Group B- Furcation Treatment with Allograft and GTR
  Interventions: Procedure: Furcation Treatment with Allograft and GTR; Device: allograft and guided tissue regeneration (GTR) membrane (DFDBM and Healiguide)

INTERVENTIONS:
Procedure: Furcation treatment with PRF — PRF Placed into the furcation after flap elevation and debridement
  Other Names: Furcation Management with Platelet rich fibrin
  Arms: 11 Patients with Grade II Manibular Molar Furcation
Procedure: Furcation Treatment with Allograft and GTR — Allograft and GTR placed into furcation after flap elevation and debridement
  Other Names: Furcation Management with DFDBM and Healiguide
  Arms: 11 Patients with Grade II Mandibular Molar Furcation D
Device: allograft and guided tissue regeneration (GTR) membrane (DFDBM and Healiguide)
  Arms: 11 Patients with Grade II Mandibular Molar Furcation D
Device: autologous platelet-rich fibrin
  Arms: 11 Patients with Grade II Manibular Molar Furcation

SUMMARY:
Background: Furcation is the bifurcation or trifurcation of a multirooted tooth. It is an area of complex anatomic morphology difficult to debride by routine periodontal instrumentation. Multiple approaches have been used in an effort to treat the furcation Choukroun's platelet-rich fibrin (PRF), a second generation platelet concentrate has biochemical components which have well known synergetic effects on healing processes. The present study was conducted to evaluate the effectiveness of autologous platelet-rich fibrin (PRF) in the treatment of mandibular molar Grade 2 furcation defects in comparison to allograft and guided tissue regeneration (GTR) membrane.

DETAILED DESCRIPTION:
ABSTRACT Background: Furcation is the bifurcation or trifurcation of a multirooted tooth. It is an area of complex anatomic morphology difficult to debride by routine periodontal instrumentation. Multiple approaches have been used in an effort to treat the furcation Choukroun's platelet-rich fibrin (PRF), a second generation platelet concentrate has biochemical components which have well known synergetic effects on healing processes. The present study was conducted to evaluate the effectiveness of autologous platelet-rich fibrin (PRF) in the treatment of mandibular molar Grade 2 furcation defects in comparison to allograft and guided tissue regeneration (GTR) membrane. MATERIALS AND METHODS: The study was designed as a randomized, prospective, parallel-arm, interventional clinical trial wherein 30 patients with periodontitis and grade II Mandibular furcation defects attending the Out Patient wing of the Department of Periodontics of a tertiary referral care hospital were equally divided into group A and group B. Patients in.Group A, were treated by the placement of PRF as a Graft and as a membrane at the surgical site , while in Group B, the defects were treated by the placement of Allograft and Healiguide collagen membrane. Plaque Index, Probing depth, Vertical clinical attachment level, Horizontal clinical attachment level, Gingival marginal level, and amount of bonefill using Radiovisiography were recorded at baseline and 9 months. Intra-group comparison of Mean scores between Group A and Group B was done using Paired t test and Inter-group comparison using independent sample t test. CONCLUSION Further studies evaluating the efficacy of PRF using a larger sample size should be performed to evaluate its true beneficial effects on long term basis in patients with mandibular molar Grade 2 furcation defects.

ELIGIBILITY:
Inclusion Criteria:

* One or more sites showing grade II furcation involvement in mandibular molars, with Probing pocket depth ≥ 5mm
* Vertical attachment level and horizontal level ≥3mm were considered.
* Patients who were systemically healthy, with no history of endodontic and periodontal treatment for the last 6 months, and no antibiotic usage for the last 6 months were included in the study. Care was taken to ascertain that the samples taken for the study were not allergic to any drugs nor to the graft materials used.

Exclusion Criteria:

* Patients with a history of diabetes, hypertension, on anticoagulant or steroid therapy (which could alter the effects of PRF), cardiac diseases, insufficient platelet counts and immunocompromised individuals were excluded from the study.
* Care was taken to exclude pregnant women and lactating mothers, smokers, patients with previous history of graft placement in the experimental site, and importantly those patients who were unable to maintain good oral hygiene (PI Score ≥ 1.5).
* If Grade II mobility was observed after phase I therapy in the experimental teeth, they were excluded

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2012-09; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Vertical clinical attacment level | 9 months Post treatment
  The Vertical clinical attachment level was assessed preoperatively and 9 months after surgery
Horizontal clinical attachment level | 9 months Post treatment
  The horizontal clinical attachment level was assessed preoperatively and 9 months after surgery.
Bone fill | 9 months Post treatment
  Bone fill was assessed radiographically and 9 months after surgery

SECONDARY OUTCOMES:
Plaque Index | 9 Months Post treatment
  Plaque index was assessed preoperatively and 9 months after surgery
Probing depth | 9 Months Post treatment
  Probing depth was assessed preoperatively and 9 months after surgery
Gingival marginal level | 9 months post treatment
  Gingival marginal level was assessed preoperatively and 9 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Rekha R Koduganti, MDS(Perio), Study Director — Prof & HOD,Dept of Periodontics,Panineeya Institute of dental sciences; Syed Asimuddin, MDS(Perio), Principal Investigator — PG Student,Panineeya Institute of Dental Sciences

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Choukroun J, Diss A, Simonpieri A, Girard MO, Schoeffler C, Dohan SL, Dohan AJ, Mouhyi J, Dohan DM. Platelet-rich fibrin (PRF): a second-generation platelet concentrate. Part IV: clinical effects on tissue healing. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2006 Mar;101(3):e56-60. doi: 10.1016/j.tripleo.2005.07.011. PMID 16504852
- [Result] Bosshardt DD, Sculean A. Does periodontal tissue regeneration really work? Periodontol 2000. 2009;51:208-19. doi: 10.1111/j.1600-0757.2009.00317.x. No abstract available. PMID 19878476
- [Result] Luepke PG, Mellonig JT, Brunsvold MA. A clinical evaluation of a bioresorbable barrier with and without decalcified freeze-dried bone allograft in the treatment of molar furcations. J Clin Periodontol. 1997 Jun;24(6):440-6. doi: 10.1111/j.1600-051x.1997.tb00209.x. PMID 9205924